CLINICAL TRIAL: NCT04094324
Title: Mental Health in Children and Youth Within Pediatric Care.
Acronym: PHU
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: HBG/MMÖ PED2019
Record Dates: First submitted 2019-04-03; First posted 2019-09-18 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Mental Health Impairment; Obesity, Adolescent; IBD
Keywords: Mental health, pediatric medicine, obesity, IBD
MeSH Terms: conditions — Pediatric Obesity; Psychological Well-Being; Obesity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children and youth at obesity clinic: Children 11-18 who are patients at obesity clinics in region Skåne SUS.
  Interventions: Behavioral: Questionnaires
- Children and youth at a pediatric gastrointestinal clinic: Children 11-18 who are patients at a gastrointestinal clinic i region Skåne SUS.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — 4 questionnaires will be answered via iPads

SUMMARY:
Over the last decades, there has been an increase in the number of children and youth with mental illness, such as anxiety and depression. Mental illness in youth has a strong negative influence on the youth's quality of life and generally leads to dysfunction in several important areas, such as school and social activities. Early detection and treatment of mental illness entails great treatment benefits, and thus provide opportunity to prevent or reduce individual suffering.

Youth who suffer från Medical conditions, such as diabetes, epilepsy, gastro-intestinal disease, and obesity, show an increased risk of developing mental illness. There are well-established, careful programs for examining somatic co-morbidities to diseases in children and youth. Currently, despite the fact that mental illness is more common in these children than medical sequelae and despite that such a procedure is recommended, no routine exist for examining mental health in children and youth presenting for treatment at pediatric clinics in Skåne. The absence of such a general screening entails that mental illness rarely is recognized by medical care providers until it has become severe.

The purpose of this study is to describe the prevalence of mental illness in children and adolescents, 11-18 years of age, that undergo Medical treatment at a Clinic for children and youth. Groups recruited for the first part of the study are obesity clinics and gastro clinics. In addition, we want to examine if mental health affects outcome success in their medical treatment. The long-term main objective of this project is early discovery and treatment of mental illness in somatically ill children and youth, thereby preventing the development of severe mental illness, and to reduce suffering.

By the end of the project we will have a well-functioning routine for examining mental health status in 11-18 years olds that present for and undergo treatment in Clinics for children and youth in Skåne. Furthermore, we hope that the screening tool can contribute to, and affect, nationally established guide-lines regarding the discovery and treatment of mental illness in children and adolescents within pediatric care.

DETAILED DESCRIPTION:
Children and youth, 11-18 years of age, that receive treatment for obesity or Irritable Bowel Disease (IBD), will be asked to fill out three questionnaires on an iPad during a regular visit at their clinic. Information about the study will be sent home before the visit, and will be repeated again at the clinic.

The questionnaires takes about 10-15 minutes in total to answer, and the Child will be able to sit in a separate room while answering. The questionnaires are well validated screening tools for various forms of mental illness; General anxiety disorder 7 item scale (GAD-7) (anxiety), Psycic Health questionnaire 8 items (PHQ-8) (depression), The Child Eating Disorder Examination 8 items (ChEDE-Q8) (eating habits), and Pediatric quality of Life inventory (PedsQL).

Patients that receive high scores will be offered a psychologist appointment for further evaluation and treatment (e. g. individual- or family centered therapy).

ELIGIBILITY:
Inclusion Criteria:

- Children and youth who are patients at a pediatric clinic in Region Skåne SUS(obesity, gatronomy)

Exclusion Criteria:

Children who are unable to reply qustions on an iPad, due to language difficulties or cognitive challenges.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and youth (11-18y) who are patients at a pediatric clinic in Region Skåne SUS (obesity, gatronomy).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Eating Disorder Examination-Questionnaire for children (ChEDE-Q8) | 2020-2022
  Self-reported eating habits Minimum maximum score: 0-6 Total: 48 Better or worse score: 0= never (no problematic eating habits) 6=daily (very problematic eating habits). High svore = very problematic eating habits
The psychic health questionnaire 8 items (PHQ-8) | 2020-2022
  Self-reported signs of depression Minimum maximum score: 0-3 Total: 24 Better or worse score: 0= never (never experiences depressive thoughts) 4=daily (experiences depressive thoughts daily). High score = high levels of depression
General anxiety scale 7 items (GAD-7) | 2020-2022
  Self-reported signs of anxiety Minimum maximum score: 0-3 Total: 21 Better or worse score: 0= never (never experiences anxiety) 4=daily (experiences anxiety daily). High score = excessive feelings of anxiety
Pediatric quality of Life scale (PedsQL) 23 items | 2020-2022
  Self-reported quality of life. Measures feelings of generel well-being Minimum maximum score: 0-4 Total: 92 Better or worse score: 0= never (never experiences well-being) 4=daily (experiences well-being daily). High score = good genereal well-being
Changes in ISO-BMI | 2021-2022
  Measures treatment outcome in obese Children by comparing ISO-BMi levels 1y apart.
Changes in F-kalprotectin levels | 2021-2022
  Measures treatment outcome in Children with iriitable bowel disease (IBD) by comparing levels 1y apart.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Helsingborgs lasarett BUM, Helsingborg
  - BÖE SUS, Malmo

IPD SHARING:
Plan to Share IPD: No